CLINICAL TRIAL: NCT03871881
Title: The Impact of Congenital Heart Disease on Neurodevelopmental Outcome and Comorbidity in Adulthood
Brief Title: Impact of Congenital Heart Disease on Neurodevelopmental Outcome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Benjamin Asschenfeldt Arlander, MD, Medical doctor, Principal investigator, University of Aarhus
Other Study IDs: Brain&CHD
Record Dates: First submitted 2017-11-22; First posted 2019-03-12 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2020-08

CONDITIONS: Heart Defects, Congenital
Keywords: Magnetic resonance imaging; Brain; Neuropsychology; Heart Defects, Congenital; Follow-Up Studies
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Magnetic Resonance Spectroscopy; Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Atrial septal defect: Patients with an open atrial septal defect, diagnosed in childhood
  Interventions: Other: Magnetic Resonance Imaging; Other: Neuropsychological assessment
- Ventricular septal defect: Patients who had surgical closure of a ventricular septal defect in childhood
  Interventions: Other: Magnetic Resonance Imaging; Other: Neuropsychological assessment
- Healthy control: Healthy, young adults matched on age, gender and education
  Interventions: Other: Magnetic Resonance Imaging; Other: Neuropsychological assessment

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Magnetic Resonance Imaging (MRI) of the brain's macro- and microstructures. Furthermore, brain regional interactions and activity is examined with quantitative functional-MRI (fMRI)
Other: Neuropsychological assessment — A special designed neuropsychological test battery of validated tests to assess function of cognitive domains

SUMMARY:
The project aims toward clarifying the underlying mechanism and the long-term impact of congenital heart disease on neurodevelopment.

DETAILED DESCRIPTION:
The project provides detailed information on the impact of congenital heart disease on neurodevelopmental outcome in adulthood. The study investigates if brain maturation and development, and the neurocognitive outcome is compromised in patients with atrial or ventricular septal defects more than 20 years after diagnosis and treatment. Data on brain morphology, brain tissue architecture, and resting-state function will be obtained by 3.0 Tesla MRI. Data on neurocognitive outcome will be obtained by a customized wide neuropsychological test battery. This study will clarify the extent of these patients' neurodevelopmental challenges and guide evaluate targeted interventions to alleviate potentially long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* ICD codes DX Q21.0 (VSD) or DX Q21.1 (ASD), surgically repaired VSD or open ASD

Exclusion Criteria:

* lack of medical record, suffering from coronary artery disease or other congenital cardiac abnormalities, diagnosed syndromes, spontaneous closure of the atrial septum defect before inclusion-date, magnetic implants or non-MRI compatible foreign objects, pregnancy, lack of Danish language skills or suffering from severe lung disease

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants are either adults who in childhood were diagnosed with an ASD or VSD, or healthy matched controls.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Long-term impact of congenital heart disease on brain development | 12 months
  MRI analysis

SECONDARY OUTCOMES:
Long-term impact of congenital heart disease on neurocognitive outcome | 12 months
  Neuropsychological assessment

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Hjortdal, MD, PhD, Study Chair — University of Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

REFERENCES:
- [Derived] Asschenfeldt B, Evald L, Salvig C, Heiberg J, Ostergaard L, Eskildsen SF, Hjortdal VE. Altered Cerebral Microstructure in Adults With Atrial Septal Defect and Ventricular Septal Defect Repaired in Childhood. J Am Heart Assoc. 2022 Jun 21;11(12):e020915. doi: 10.1161/JAHA.121.020915. Epub 2022 Jun 14. PMID 35699183
- [Derived] Lau-Jensen SH, Asschenfeldt B, Evald L, Hjortdal VE. Hyperactivity and Inattention in Young Patients Born With an Atrial Septal or Ventricular Septal Defect. Front Pediatr. 2021 Dec 6;9:786638. doi: 10.3389/fped.2021.786638. eCollection 2021. PMID 34938699
- [Derived] Asschenfeldt B, Evald L, Yun HJ, Heiberg J, Ostergaard L, Grant PE, Hjortdal VE, Im K, Eskildsen SF. Abnormal Left-Hemispheric Sulcal Patterns in Adults With Simple Congenital Heart Defects Repaired in Childhood. J Am Heart Assoc. 2021 Apr 6;10(7):e018580. doi: 10.1161/JAHA.120.018580. Epub 2021 Mar 22. PMID 33745293
- [Derived] Asschenfeldt B, Evald L, Heiberg J, Salvig C, Ostergaard L, Dalby RB, Eskildsen SF, Hjortdal VE. Neuropsychological Status and Structural Brain Imaging in Adults With Simple Congenital Heart Defects Closed in Childhood. J Am Heart Assoc. 2020 Jun 2;9(11):e015843. doi: 10.1161/JAHA.120.015843. Epub 2020 May 19. PMID 32427039